CLINICAL TRIAL: NCT00560209
Title: Study of ONO-1101 in Patients Scheduled for Coronary Angiography, a Double-Blind, Randomized,Placebo-Controlled, Parallel Group, Multi-Center Study
Brief Title: Study of ONO-1101 in Patients Scheduled for Coronary Angiography
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ONO-1101-26
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Artery Disease
Keywords: ONO-1101; Coronary Artery Disease; Multi-slice CT
MeSH Terms: conditions — Coronary Artery Disease | interventions — landiolol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- P (Placebo Comparator)
  Interventions: Drug: ONO-1101
- E2 (Experimental)
  Interventions: Drug: ONO-1101
- E1 (Experimental)
  Interventions: Drug: ONO-1101

INTERVENTIONS:
Drug: ONO-1101 — placebo for 1 minute IV
  Arms: P
Drug: ONO-1101 — 0.06 mg/kg for 1 minute IV
  Arms: E1
Drug: ONO-1101 — 0.125 mg/kg for 1 minute IV
  Arms: E2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ONO-1101 in patients scheduled for coronary angiography, in a double-blind, randomized, placebo-controlled, parallel group, multi-center study.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older
* Heart rate less than 90 beats/min and more than 70 beats/min at entering the CT room

Exclusion Criteria:

* Previous allergic reactions to contrast agent
* Renal failure
* Asthma
* Concomitant beta-receptor blocking agent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
CT image quality | one day

SECONDARY OUTCOMES:
Heart rate | For less than one month
CT diagnostic accuracy | For less than one month

CONTACTS AND LOCATIONS:
Overall Officials: Shinichi Kikawa, Study Director — Ono Pharmaceutial Co., Ltd
Locations (1):
- Kinki Region, Kinki, Japan

REFERENCES:
- [Derived] Jinzaki M, Hirano M, Hara K, Suzuki T, Yamashina A, Ikari Y, Iino M, Yamaguchi T, Kuribayashi S. A randomized, double-blind, placebo-controlled, phase II dose-finding study of the short acting beta1-blocker, landiolol hydrochloride, in patients with suspected ischemic cardiac disease. Int J Cardiovasc Imaging. 2013 Jun;29 Suppl 1(Suppl 1):7-20. doi: 10.1007/s10554-013-0253-3. Epub 2013 Jun 20. PMID 23784548